CLINICAL TRIAL: NCT06456723
Title: Evaluation of [18F]Fluoroethyl Triazole Labelled [Tyr3]-Octreotate Analogues for the Imaging of Neuroendocrine Tumours.
Acronym: FETONET
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Imperial College Healthcare NHS Trust (Other); Royal Marsden NHS Foundation Trust (Other); University of Manchester (Other); The Christie NHS Foundation Trust (Other); Invicro (Other); Newcastle University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 13HH0807
Record Dates: First submitted 2024-05-28; First posted 2024-06-13 (Actual); Results first posted 2025-05-01 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Neuroendocrine Tumors
Keywords: Positron Emission Tomography
MeSH Terms: conditions — Neuroendocrine Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part A: [18F]-FET-βAG-TOCA-PET/CT performed in patients with histologically-confirmed NET. (Experimental): Patients with histologically-confirmed neuroendocrine tumours (NET) enrolled into Part A of the FETONET study underwent whole-body dynamic [18F]FET-βAG-TOCA imaging at multiple time points over a 4 hour period, with sampling of venous bloods for radioactivity and radioactive metabolite quantification.
  Interventions: Drug: [18F]-FET-βAG-TOCA
- Part B: [18F]FET-βAG-TOCA PET/CT compared with [68Ga]Ga-DOTA-peptide PET/CT in patients with NET. (Experimental): Patients with histologically confirmed neuroendocrine tumours (NET) underwent PET/CT imaging with both [18F]FET-βAG-TOCA and [68Ga]Ga-DOTA-peptide. The two PET/CT scans were performed within a 6-month time period. Whole-body static [18F]FET-βAG-TOCA PET/CT scan performed at 50 minutes post radiotracer injection.
  Interventions: Drug: [18F]-FET-βAG-TOCA

INTERVENTIONS:
Drug: [18F]-FET-βAG-TOCA — Single I.V. administration of a [18F]fluoroethyl triazole [Tyr3]Octreotate ([18F]-FET-βAG-TOCA). Patients will receive a maximum injected dose of 370MBq and will subsequently undergo PET/CT imaging.

SUMMARY:
Radiolabelled somatostatin analogs are invaluable in the diagnosis and treatment of neuroendocrine tumours (NET). The most common positron emission tomography (PET) radiotracers used for the visualisation of NET are radiolabelled somatostatin analogs (SSAs) labelled with [68Ga]Ga-DOTA-peptides. However, [68Ga]Ga-DOTA-peptide radiolabelled SSAs have significant limitations in terms of accessibility and low throughput. The team at Imperial College London developed a novel radiotracer, [18F]fluoroethyl triazole labelled [Tyr3]-Octreotate analogue ([18F]-FET-βAG-TOCA), in an attempt to overcome these limitations. The FETONET study was designed to have 3 parts. The FETONET study was designed to have 3 parts. Part A evaluated the biodistribution, dosimetry and safety of [18F]FET-βAG-TOCA. Uptake was assessed at multiple time points over a 4 hour period. The data was analysed and an optimal imaging time point determined. Part B of the FETONET study involved the performance of whole body static [18F]FET-βAG-TOCA PET-CT imaging, at the optimal time point previously established, within a larger cohort of patients. Part C comprised a prospective non-inferiority study that analysed the [18F]FET-βAG-TOCA PET/CT data collected within Part A & Part B and compared this to standard of care [Ga68]Ga-DOTA-peptide PET-CT imaging.

DETAILED DESCRIPTION:
Neuroendocrine tumours (NET) are tumours derived from enterochromaffin cells, which are characterised by the expression of somatostatin receptors (SSTRs) on their surface. These tumours release substances into systemic circulation, resulting in episodic flushing, wheezing, diarrhoea, and eventual right-sided valvular heart disease. All of these symptoms negatively impact on patients' quality of life. The management of NET is primarily determined by the stage of disease. For patients with localised or limited disease the primary modality of therapy is surgery. Whilst patients with metastatic disease, undergo systemic therapy with palliative intent. Accurate imaging is therefore central to the management of this disease. Whilst computed tomography (CT) is useful in the localisation of NET, nuclear imaging using tumour-specific radiolabelled receptors are considerably more sensitive and specific methods for detecting NET and their metastases. The most commonly used positron emission tomography (PET) radiotracers used for the visualisation of NET are radiolabelled somatostatin analogs (SSAs) labelled with [68Ga]Ga-DOTA-peptides. The [68Ga]Ga-DOTA-peptide radiolabelled SSAs have significant limitations in terms of accessibility and low throughput. The team at Imperial College London developed a novel radiotracer, [18F]fluoroethyl triazole labelled [Tyr3]-Octreotate analogue ([18F]-FET-βAG-TOCA), in an attempt to overcome these limitations. The FETONET study was designed to have 3 parts. The FETONET study was designed to have 3 parts. Part A evaluated the biodistribution, dosimetry and safety of [18F]FET-βAG-TOCA. Uptake was assessed at multiple time points over a 4 hour period. The data was analysed and an optimal imaging time point determined. Part B of the FETONET study involved the performance of whole body static [18F]FET-βAG-TOCA PET-CT imaging, at the optimal time point previously established, within a larger cohort of patients. Part C comprised a prospective non-inferiority study that analysed the [18F]FET-βAG-TOCA PET/CT data collected within Part A & Part B and compared this to standard of care [Ga68]Ga-DOTA-peptide PET-CT imaging.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Age ≥ 18 years
* Histological diagnosis of NET of any site, except where ENETS criteria does not mandate histology for confirmation of diagnosis or patients who have a positive 68Gallium-peptide scan in whom NET diagnosis is pre-operatively definitive.
* Locally advanced or metastatic disease.
* Eastern Cooperative Oncology Group (ECOG) performance status of <2 (appendix A).
* Life expectancy > 3 months.
* Measurable disease defined as a lesion that can be accurately measured in at least one dimension with the longest diameter ≥10mm using conventional techniques.
* Somatostatin receptor imaging within 6 months. (if patient does not have somatostatin receptor imaging they may also be included provided they have measurable disease (≥10mm) on conventional imaging.
* Adequate organ system function as defined within Table 1.

Exclusion Criteria:

* Patients received chemotherapy within 3 weeks of study.
* Patients received radiotherapy within 4 weeks of study.
* Active uncontrolled infections, gastrointestinal disease, haemolysis or any serious co-existing medical illness.
* Psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule.
* Pregnant or lactating women.
* Females of childbearing potential who are unwilling to avoid pregnancy, for the duration of the study.
* Presence of any underlying medical conditions which in the investigators opinion would make the patients unsuitable for treatment.
* Patient not expected to be able to tolerate the scanning sessions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2014-05-14 (Actual); Primary Completion 2018-10-17 (Actual); Study Completion 2018-10-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rohini Sharma, Study Chair — Imperial College London

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers.

REFERENCES:
- [Background] Dubash SR, Keat N, Mapelli P, Twyman F, Carroll L, Kozlowski K, Al-Nahhas A, Saleem A, Huiban M, Janisch R, Frilling A, Sharma R, Aboagye EO. Clinical Translation of a Click-Labeled 18F-Octreotate Radioligand for Imaging Neuroendocrine Tumors. J Nucl Med. 2016 Aug;57(8):1207-13. doi: 10.2967/jnumed.115.169532. Epub 2016 May 12. PMID 27173162
- [Result] Dubash S, Barwick TD, Kozlowski K, Rockall AG, Khan S, Khan S, Yusuf S, Lamarca A, Valle JW, Hubner RA, McNamara MG, Frilling A, Tan T, Wernig F, Todd J, Meeran K, Pratap B, Azeem S, Huiban M, Keat N, Lozano-Kuehne JP, Aboagye EO, Sharma R. Somatostatin Receptor Imaging with [18F]FET-betaAG-TOCA PET/CT and [68Ga]Ga-DOTA-Peptide PET/CT in Patients with Neuroendocrine Tumors: A Prospective, Phase 2 Comparative Study. J Nucl Med. 2024 Feb 8;65(3):416-22. doi: 10.2967/jnumed.123.266601. Online ahead of print. PMID 38331457

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: 14May2014-17Oct2018. The FETONET study was designed to have 3 parts. Part A evaluated the biodistribution, dosimetry and safety of [18F]FET-βAG-TOCA. Uptake was assessed at multiple time points and an optimal time point determined. Part B utilised this time point within a larger cohort. Part C comprised a prospective non-inferiority study analysing the [18F]FET-βAG-TOCA PET/CT data collected during Parts A & B and comparing this to [Ga68]Ga-DOTA-peptide PET-CT imaging.
Groups:
- Part A: [18F]-FET-βAG-TOCA-PET/CT Performed in Patients With Histologically-confirmed NET.: Patients with histologically-confirmed neuroendocrine tumours (NET) enrolled into Part A of the FETONET study underwent whole-body dynamic [18F]-FET-βAG-TOCA PET/CT imaging at multiple time points over a 4 hour period, with sampling of venous bloods for radioactivity and radioactive metabolite quantification.
  The maximum dose of [18F]-FET-βAG-TOCA injected was 165MBq.
  Imaging Protocol for patients in Part A of the FETONET study:
  -2 minutes - Low dose attenuation CT.
  0 minutes - Injection of [18F]-FET-βAG-TOCA (maximum of 165MBq)
  0-242 - Dynamic whole body [18F]-FET-βAG-TOCA PET-CT (6 sweeps of the body). Following the fourth sweep, the patient had a 20 minutes break. The patient returned to the PET-CT scanner and had a second low-dose attenuation CT scan before completing PET/CT sweeps 5 & 6.
  Total effective dose: 12 mSv
  In Part A of the FETONET study, two low-dose attenuation CT scans were performed per patient. Whereas, only one low-dose attenuation CT scan was performed per patient in Part A. The total effective dose per patient was therefore higher in Part A.
- Part B: [18F]-FET-βAG-TOCA-PET/CT Compared With [68Ga]Ga-DOTA-peptide PET/CT in Patients With NET.: Patients with histologically confirmed neuroendocrine tumours (NET) underwent PET/CT imaging with both [18F]-FET-βAG-TOCA and [68Ga]Ga-peptide. The two PET/CT scans were performed within a 6-month time period.
  Whole-body static [18F]-FET-βAG-TOCA PET-CT imaging was conducted 50 minutes post-injection.
  The maximum dose of [18F]-FET-βAG-TOCA injected was 165MBq.
  Imaging Protocol for patients in Part B of the FETONET study:
  -2 minutes - Low dose attenuation CT.
  0 minutes - Injection of the [18F]-FET-βAG-TOCA (Maximum injected dose of 370MBq)
  * 50 minutes - [18F]-FET-βAG-TOCA PET scan 1
  * 120 minutes - [18F]-FET-βAG-TOCA PET scan 2
  Total effective dose: 9 mSv
  In Part B of the FETONET study, one low-dose attenuation CT scan was performed per patient. Whereas, two low-dose attenuation CT scans were performed per patient in Part A. The total effective dose per patient was therefore lower in Part B.
Period: Part A
Arm/Group | Part A: [18F]-FET-βAG-TOCA-PET/CT Performed in Patients With Histologically-confirmed NET. | Part B: [18F]-FET-βAG-TOCA-PET/CT Compared With [68Ga]Ga-DOTA-peptide PET/CT in Patients With NET.
Started | 9 | 0
Completed (Part A - A first-in-human study to evaluate the biodistribution, dosimetry and safety of [18F]FET-βAG-TOCA in patients with histologically-confirmed NET. [18F]FET-βAG-TOCA uptake was evaluated at multiple time points over a period of 4 hours to allow for the determination of an optimal time point.) | 9 | 0
Not Completed | 0 | 0
Period: Part B
Arm/Group | Part A: [18F]-FET-βAG-TOCA-PET/CT Performed in Patients With Histologically-confirmed NET. | Part B: [18F]-FET-βAG-TOCA-PET/CT Compared With [68Ga]Ga-DOTA-peptide PET/CT in Patients With NET.
Started | 0 | 47
Completed (Part B - Comparison of [18F]FET-βAG-TOCA PET/CT imaging, performed at the optimal timepoint established in Part A, against standard-of-care [68Ga]Ga-DOTA-peptide PET/CT imaging.) | 0 | 47
Not Completed | 0 | 0
Period: Part C - Primary Analysis
Arm/Group | Part A: [18F]-FET-βAG-TOCA-PET/CT Performed in Patients With Histologically-confirmed NET. | Part B: [18F]-FET-βAG-TOCA-PET/CT Compared With [68Ga]Ga-DOTA-peptide PET/CT in Patients With NET.
Started | 9 | 47
Completed (Part C - A prospective non-inferiority study comparing [18F]FET-βAG-TOCA PET/CT imaging, performed at the optimal timepoint, against SoC [68Ga]Ga-DOTA-peptide PET/CT . Part C of the FETONET study comprised a prospective non-inferiority study comparing the [18F]FET-βAG-TOCA PET/CT and [68Ga]Ga-DOTA-peptide PET/CT data collected from patients enrolled in Part A and Part B.) | 9 | 36
Not Completed | 0 | 11

BASELINE CHARACTERISTICS:
Population: The FETONET study was designed to have 3 parts. Part A evaluated the biodistribution, dosimetry and safety of [18F]FET-βAG-TOCA. Radiotracer uptake was assessed at multiple time points over 4 hours. An optimal imaging time point was determined. Part B utilised this time point within a larger cohort. Part C comprised a prospective non-inferiority study, analysing the [18F]FET-βAG-TOCA PET/CT data collected during Parts A & B, and comparing this to [Ga68]Ga-DOTA-peptide PET-CT imaging (SoC).
Groups:
- Part A: [18F]-FET-βAG-TOCA-PET/CT Performed in Patients With Histologically-confirmed NET.: Patients with histologically confirmed neuroendocrine tumours (NET) enrolled into Part A of the FETONET study underwent whole-body dynamic [18F]-FET-βAG-TOCA PET/CT imaging at multiple time points over a 4-hour period, with sampling of venous bloods for radioactivity and radioactive metabolite quantification.
  The maximum dose of [18F]-FET-βAG-TOCA injected was 165MBq.
  Imaging Protocol for patients in Part A of the FETONET study:
  -2 minutes - Low dose attenuation CT.
  0 minutes - Injection of [18F]-FET-βAG-TOCA (maximum of 165MBq)
  0-242 - Dynamic whole body [18F]-FET-βAG-TOCA PET-CT (6 sweeps of the body). Following the fourth sweep, the patient had a 20 minutes break. The patient returned to the PET-CT scanner and had a second low-dose attenuation CT scan before completing PET/CT sweeps 5 & 6.
  Total effective dose: 12 mSv
  In Part A of the FETONET study, two low-dose attenuation CT scans were performed per patient. Whereas, only one low-dose attenuation CT scan was performed per patient in Part A. The total effective dose per patient was therefore higher in Part A.
- Total: Total of all reporting groups
Arm/Group | Part A: [18F]-FET-βAG-TOCA-PET/CT Performed in Patients With Histologically-confirmed NET. | Part B: [18F]-FET-βAG-TOCA-PET/CT Compared With [68Ga]Ga-DOTA-peptide PET/CT in Patients With NET. | Total
Number analyzed (Participants) | 9 | 36 | 45
Age, Continuous [Median (Full Range); unit: years] | 56 [35 to 73] | 60.5 [29 to 81] | 57 [29 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 16 | 22
  Male | 3 | 20 | 23
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Site of Primary Tumour [Count of Participants; unit: Participants]
  Pancreas | 3 | 12 | 15
  Small Bowel | 3 | 17 | 20
  Lung | 3 | 0 | 3
  Other | 0 | 7 | 7
Tumour Grade - Histological Confirmation [Count of Participants; unit: Participants] — Histological confirmation of tumour grade. Grade 1 NETs consist of cells that look very similar to normal cells. Tumours are slow growing and less likely to spread - well differentiated tumours.
  Grade 2 NETs consist of cells that look less like normal cells and are more likely to grow and spread - moderately differentiated tumours.
  Participants
    Grade 1 | 2 | 13 | 15
    Grade 2 | 7 | 14 | 21
    Unknown | 0 | 9 | 9

OUTCOME MEASURES:

1. Primary Outcome: To Determine the Biodistribution of [18F] Following Single I.V Administration of [18F]-FET-βAG-TOCA Injection in Patients With a Histological Diagnosis of NET.
Description: Mean residence time (MRT) was used to characterise the biodistribution of [18F]-FET-βAG-TOCA throughout the body. Mean residence time is a pharmacokinetic/uptake parameter that describes the average length of time a radiotracer resides within the body, or a particular organ, before being eliminated. Understanding MRT helps researchers to determine how long a radiotracer remains in the system, which is crucial for drug dosing, therapeutic efficacy, and potential toxicity assessment.
Time Frame: Baseline (on day of scan over 4 hours)
Population: The number of participants analysed differ within certain rows (breasts, ovaries, uterus and testes due to the anatomical differences between the participant groups.
Measure: Mean (Standard Deviation); unit: Mean Residence Time (MBq-h/MBq)
Groups:
- Part A: [18F]-FET-βAG-TOCA-PET/CT Performed in Male Patients With Histologically-confirmed NET.: Mean residence time (MBq.h/MBq) of [18F]-FET-βAG-TOCA within the organs of the male participants enrolled into Part A of the FETONET study.
  Patients with histologically confirmed neuroendocrine tumours (NET) enrolled into Part A of the FETONET study underwent whole-body dynamic [18F]-FET-βAG-TOCA PET/CT imaging at multiple time points over a 4-hour period, with sampling of venous bloods for radioactivity and radioactive metabolite quantification.
  The maximum dose of [18F]-FET-βAG-TOCA injected was 165MBq.
  Imaging Protocol for patients in Part A of the FETONET study:
  -2 minutes - Low dose attenuation CT.
  0 minutes - Injection of [18F]-FET-βAG-TOCA (maximum of 165MBq)
  0-242 - Dynamic whole body [18F]-FET-βAG-TOCA PET-CT (6 sweeps of the body). Following the fourth sweep, the patient had a 20 minutes break. The patient returned to the PET-CT scanner and had a second low-dose attenuation CT scan before completing PET/CT sweeps 5 & 6.
  Total effective dose: 12 mSv
  In Part A of the FETONET study, two low-dose attenuation CT scans were performed per patient. Whereas, only one low-dose attenuation CT scan was performed per patient in Part A. The total effective dose per patient was therefore higher in Part A.
- Part A: [18F]-FET-βAG-TOCA-PET/CT Performed in Female Patients With Histologically-confirmed NET.: Mean residence time (MBq.h/MBq) of [18F]-FET-βAG-TOCA within the organs of the female participants enrolled into Part A of the FETONET study.
  Patients with histologically confirmed neuroendocrine tumours (NET) enrolled into Part A of the FETONET study underwent whole-body dynamic [18F]-FET-βAG-TOCA PET/CT imaging at multiple time points over a 4-hour period, with sampling of venous bloods for radioactivity and radioactive metabolite quantification.
  The maximum dose of [18F]-FET-βAG-TOCA injected was 165MBq.
  Imaging Protocol for patients in Part A of the FETONET study:
  -2 minutes - Low dose attenuation CT.
  0 minutes - Injection of [18F]-FET-βAG-TOCA (maximum of 165MBq)
  0-242 - Dynamic whole body [18F]-FET-βAG-TOCA PET-CT (6 sweeps of the body). Following the fourth sweep, the patient had a 20 minutes break. The patient returned to the PET-CT scanner and had a second low-dose attenuation CT scan before completing PET/CT sweeps 5 & 6.
  Total effective dose: 12 mSv
  In Part A of the FETONET study, two low-dose attenuation CT scans were performed per patient. Whereas, only one low-dose attenuation CT scan was performed per patient in Part A. The total effective dose per patient was therefore higher in Part A.
Arm/Group | Part A: [18F]-FET-βAG-TOCA-PET/CT Performed in Male Patients With Histologically-confirmed NET. | Part A: [18F]-FET-βAG-TOCA-PET/CT Performed in Female Patients With Histologically-confirmed NET.
Number analyzed (Participants) | 3 | 6
Mean Residence Time (MBq-h/MBq)
  Adrenals | 0.002 (0.0002) | 0.003 (0.0008)
  Brain | 0.006 (0.001) | 0.007 (0.001)
  Breasts: number analyzed (Participants) | 0 | 6
  Breasts |  | 0.004 (0.001)
  Cortical Bone | 0.049 (0.002) | 0.040 (0.016)
  Gallbladder: number analyzed (Participants) | 1 | 6
  Gallbladder | 0.110 | 0.072 (0.019)
  Heart Contents | 0.029 (0.014) | 0.019 (0.005)
  Heart Wall | 0.020 (0.010) | 0.013 (0.004)
  Kidneys | 0.088 (0.007) | 0.089 (0.026)
  Liver | 0.478 (0.073) | 0.089 (0.084)
  Lungs | 0.063 (0.009) | 0.067 (0.025)
  Lower Large Intestine | 0.012 (0.002) | 0.019 (0.011)
  Muscle | 0.709 (0.154) | 0.600 (0.154)
  Ovaries: number analyzed (Participants) | 0 | 6
  Ovaries |  | 0.0005 (0.00004)
  Pancreas | 0.017 (0.006) | 0.010 (0.0035)
  Red Marrow | 0.028 (0.004) | 0.050 (0.032)
  Small Intestine | 0.094 (0.065) | 0.121 (0.055)
  Stomach | 0.005 (0.029) | 0.066 (0.222)
  Spleen | 0.122 (0.019) | 0.097 (0.026)
  Testes: number analyzed (Participants) | 3 | 0
  Testes | 0.001 (0.0002) |
  Thyroid | 0.001 (0.0003) | 0.0008 (0.0003)
  Upper Large Intestine | 0.026 (0.004) | 0.028 (0.014)
  Urinary Bladder | 0.075 (0.019) | 0.101 (0.028)
  Uterus: number analyzed (Participants) | 0 | 6
  Uterus |  | 0.006 (0.001)
  Remainder | 0.523 (0.250) | 0.628 (0.025)

2. Primary Outcome: To Calculate the Effective Dose (ED) of [18F]-FET-βAG-TOCA
Description: Effective dose is an estimate of the overall risk of potential harm from exposure to ionising radiation. ED takes into account, the absorbed dose to all organs of the body, the relative harm level of the radiation and the sensitivities of each organ to radiation. ED may help in understanding the risk of potential long-term health effects from radiation exposure, such as the risk of developing cancer later in life. The unit of measure for ED is millisievert per megabecquerel (mSv/MBq), which refers to the effective dose (amount of radiation absorbed by the body) per unit of activity administered.
Time Frame: Baseline (on the day of the scan over 4 hours)
Population: Effective dose (ED) of [18F]-FET-βAG-TOCA in patients with histologically confirmed NETs.
Measure: Mean (Standard Deviation); unit: Effective Dose (mSv/MBq)
Groups:
- Part A: [18F]-FET-βAG-TOCA-PET/CT Performed in Patients With Histologically-confirmed NET.: Effective Dose (ED) calculation for [18F]-FET-βAG-TOCA in participants with histologically confirmed neuroendocrine tumours enrolled into Part A of the FETONET study.
  Patients with histologically confirmed neuroendocrine tumours (NET) enrolled into Part A of the FETONET study underwent whole-body dynamic [18F]-FET-βAG-TOCA PET/CT imaging at multiple time points over a 4-hour period, with sampling of venous bloods for radioactivity and radioactive metabolite quantification.
  The maximum dose of [18F]-FET-βAG-TOCA injected was 165MBq.
  Imaging Protocol for patients in Part A of the FETONET study:
  -2 minutes - Low dose attenuation CT.
  0 minutes - Injection of [18F]-FET-βAG-TOCA (maximum of 165MBq)
  0-242 - Dynamic whole body [18F]-FET-βAG-TOCA PET-CT (6 sweeps of the body). Following the fourth sweep, the patient had a 20 minutes break. The patient returned to the PET-CT scanner and had a second low-dose attenuation CT scan before completing PET/CT sweeps 5 & 6.
  Total effective dose: 12 mSv
  In Part A of the FETONET study, two low-dose attenuation CT scans were performed per patient. Whereas, only one low-dose attenuation CT scan was performed per patient in Part A. The total effective dose per patient was therefore higher in Part A.
Arm/Group | Part A: [18F]-FET-βAG-TOCA-PET/CT Performed in Patients With Histologically-confirmed NET.
Number analyzed (Participants) | 9
Effective Dose (mSv/MBq) | 0.029 (0.004)

3. Primary Outcome: To Assess Tumoural Uptake of [18F]-FET-βAG-TOCA
Description: Standardised uptake value (SUV) is a semiquantitative measurement of radiotracer uptake in tissue. It is a ratio that compares the activity concentration in a specific region of interest to the activity concentration in the whole body. SUVmax is the highest value of the SUV measured within a region of interest.
Time Frame: Baseline (on the scan day over 4 hours)
Population: The FETONET study was designed to have 3 parts. Part C comprised a prospective non-inferiority study, combining the [18F]FET-βAG-TOCA PET/CT data (collected at the optimal time point) for participants enrolled into Part A and Part B and compared this to standard of care [68Ga]Ga-DOTA-peptide PET/CT imaging. This trial design was a prospective decision for the purposes of efficiency. A total of 285 lesions were detected within the 45 patients analysed using this imaging modality.
Measure: Median (Full Range); unit: SUVmax
Units Other Than Participants: Lesions
Groups:
- Part C - Primary Analysis Cohort: A prospective decision was made that the FETONET study would be comprised of 3 parts for efficiency. Part A evaluated [18F]FET-βAG-TOCA uptake at multiple time points over a 4 hour period. An optimal imaging time point was subsequently determined. Part B utilised this optimal time point within a larger cohort of patients with NET. The trial was designed in such a way that the timepoint used in Part B was congruent with one of the time points assessed in Part A. This design was was chosen to ensure efficiency in an otherwise no benefit trial for patients, which typically have a poorer recruitment rate. Part C comprised a prospective non-inferiority study, combining the [18F]FET-βAG-TOCA PET/CT data collected at the optimal time point for participants enrolled into Part A and Part B and compared this to standard of care [68Ga]Ga-DOTA-peptide PET/CT imaging.
Arm/Group | Part C - Primary Analysis Cohort
Number analyzed (Participants) | 45
Number analyzed (Lesions) | 285
SUVmax
  Head & Neck: number analyzed (Participants) | 3
  Head & Neck: number analyzed (Lesions) | 3
  Head & Neck | 12.4 [10.4 to 27.7]
  Liver: number analyzed (Participants) | 27
  Liver: number analyzed (Lesions) | 110
  Liver | 19.6 [7.2 to 132.4]
  Bone: number analyzed (Participants) | 12
  Bone: number analyzed (Lesions) | 49
  Bone | 9.7 [2.2 to 37.0]
  Pancreas: number analyzed (Participants) | 14
  Pancreas: number analyzed (Lesions) | 28
  Pancreas | 24.5 [4.2 to 85.8]
  Abdomen/Pelvis: number analyzed (Participants) | 18
  Abdomen/Pelvis: number analyzed (Lesions) | 36
  Abdomen/Pelvis | 18.8 [2.7 to 152.3]
  Lymph Nodes: number analyzed (Participants) | 10
  Lymph Nodes: number analyzed (Lesions) | 48
  Lymph Nodes | 18.0 [3.4 to 102.4]
  Lung: number analyzed (Participants) | 19
  Lung: number analyzed (Lesions) | 11
  Lung | 10.4 [5.3 to 42.1]

4. Secondary Outcome: To Compare the Diagnostic Efficacy of [18F]-FET-βAG-TOCA PET/CT With Standard of Care Somatostatin Receptor Imaging in Patients With a Histological Diagnosis of NET.
Description: To determine the clinical utility of [18F]-FET-βAG-TOCA-PET/CT compared with standard of care [68Ga]Ga-DOTA-peptide imaging. Standardised uptake value (SUV) is a semiquantitative measurement of radiotracer uptake in tissue. It is a ratio that compares the activity concentration in a specific region of interest to the activity concentration in the whole body. SUVmax is the highest value of the SUV measured within a region of interest. The median SUVmax of [18F]-FET-βAG-TOCA and [68Ga]-DOTA-peptide per anatomic region were calculated to determine diagnostic efficacy. Diagnostic efficacy is the ability of a test to correctly identify a disease or condition when it's present and correctly identify the absence of a disease when it's not present.
Time Frame: [68Ga]Ga-DOTA-peptide PET/CT imaging performed within 6 months of the [18F]-FET-βAG-TOCA PET/CT scan.
Population: The FETONET study was designed to have 3 parts. Part C comprised a prospective non-inferiority study. [18F]FET-βAG-TOCA PET/CT data collected for patients enrolled into Parts A and B of the FETONET study were combined and compared to [68Ga]Ga-DOTA-peptide PET/CT (standard of care) imaging. This trial design was a prospective decision for the purposes of efficiency. A total of 285 lesions (45 patients) were detected using [18F]-FET-βAG-TOCA & [68Ga]Ga-DOTA-peptide PET/CT imaging.
Measure: Median (Full Range); unit: Median Tumour Uptake (SUVmax)
Units Other Than Participants: Lesions
Groups:
- Part C - [18F]-FET-βAG-TOCA PET/CT; Part C - [68Ga]Ga-DOTA-peptide PET/CT: A prospective decision was made that the FETONET study would be comprised of 3 parts for efficiency. Part A evaluated [18F]FET-βAG-TOCA uptake at multiple time points over a 4 hour period. An optimal imaging time point was subsequently determined. Part B utilised this optimal time point within a larger cohort of patients with NET. The trial was designed in such a way that the time point utilised in Part B would be congruent with one of the time points assessed in Part A. This design was was chosen to ensure efficiency in an otherwise no benefit trial for patients, which typically have a poorer recruitment rate. Part C comprised a prospective non-inferiority study. [18F]FET-βAG-TOCA PET/CT data for participants enrolled into Part A and Part B (collected at the optimal imaging time point) were combined, analysed and compared to [68Ga]Ga-DOTA-peptide PET/CT data (standard of care).
Arm/Group | Part C - [18F]-FET-βAG-TOCA PET/CT | Part C - [68Ga]Ga-DOTA-peptide PET/CT
Number analyzed (Participants) | 45 | 45
Number analyzed (Lesions) | 285 | 285
Median Tumour Uptake (SUVmax)
  Head & Neck: number analyzed (Participants) | 3 | 3
  Head & Neck: number analyzed (Lesions) | 3 | 3
  Head & Neck | 12.4 [10.4 to 27.7] | 6.9 [6.4 to 23.4]
  Liver: number analyzed (Participants) | 27 | 27
  Liver: number analyzed (Lesions) | 110 | 110
  Liver | 19.6 [7.2 to 132.4] | 20.6 [6.7 to 95.1]
  Bone: number analyzed (Participants) | 12 | 12
  Bone: number analyzed (Lesions) | 49 | 49
  Bone | 9.7 [2.2 to 37.0] | 7.2 [1.9 to 38.8]
  Pancreas: number analyzed (Participants) | 14 | 14
  Pancreas: number analyzed (Lesions) | 28 | 28
  Pancreas | 24.5 [4.2 to 85.8] | 21.9 [6.4 to 88.4]
  Abdomen/Pelvis: number analyzed (Participants) | 18 | 18
  Abdomen/Pelvis: number analyzed (Lesions) | 36 | 36
  Abdomen/Pelvis | 18.8 [2.7 to 152.3] | 21.2 [4.1 to 110.3]
  Lymph Nodes: number analyzed (Participants) | 10 | 10
  Lymph Nodes: number analyzed (Lesions) | 48 | 48
  Lymph Nodes | 18.0 [3.4 to 102.4] | 17.0 [3.1 to 122.9]
  Lung: number analyzed (Participants) | 19 | 19
  Lung: number analyzed (Lesions) | 11 | 11
  Lung | 10.4 [5.3 to 42.1] | 9.4 [2.2 to 38.0]

5. Secondary Outcome: Comparison of [18F]-FET-βAG-TOCA PET/CT Scan and Central Review (Nuclear Medicine and Radiology Physician Experts) of All Imaging Received.
Description: The [18F]FET-βAG-TOCA and [68Ga]Ga-DOTA-peptide PET/CT scans were reviewed by independent imaging experts to obtain an objective inter-reader lesion detection rate. To avoid recall bias, the [18F]FET-βAG-TOCA and [68Ga]Ga-DOTA-peptide PET/CT scans for each subject were reviewed at less 4 weeks apart in random order Percentage of agreement, also known as percent agreement, is a simple method to measure inter-rater reliability (IRR), calculating the proportion of times raters agree without considering chance. It's calculated by dividing the number of agreements by the total number of ratings and multiplying by 100
Time Frame: [68Ga]Ga-DOTA-peptide PET/CT imaging assessed within 6 months of the [18F]-FET-βAG-TOCA PET/CT scan.
Population: The FETONET study was designed to have 3 parts. Part C comprised a prospective non-inferiority study. [18F]FET-βAG-TOCA PET/CT data for the patients enrolled into Parts A and B of the FETONET study (45 patients) were compared to standard of care [68Ga]Ga-DOTA-peptide PET/CT imaging. This trial design was a prospective decision for the purposes of efficiency. All PET/CT scans analysed within Part C were reviewed by independent imaging experts to determine an inter-reader lesion detection rate.
Measure: Number; unit: Percentage of Agreement
Groups:
- Part C - Inter-rater Agreement for 18F-FET-βAG-TOCA Per Anatomic Region Between All 4 Raters.: Inter-rater agreement for [18F]FET-βAG-TOCA per anatomic region between all four raters.
  All participant data analysed within Part C of the FETONET study had a [18F]FET-βAG-TOCA PET/CT scan performed at the optimal time point established following the completion of Part A and a [68Ga]Ga-DOTA-peptide PET/CT scan as per standard of care.
- Part C - Inter-rater Agreement for [68Ga]Ga-DOTA-peptide Per Anatomic Region Between All 4 Raters: Inter-rater agreement for [68Ga]Ga-DOTA-peptide per anatomic region between all four raters.
  All participant data analysed within Part C of the FETONET study had a [18F]FET-βAG-TOCA PET/CT scan performed at the optimal time point established following the completion of Part A and a [68Ga]Ga-DOTA-peptide PET/CT scan as per standard of care.
Arm/Group | Part C - Inter-rater Agreement for 18F-FET-βAG-TOCA Per Anatomic Region Between All 4 Raters. | Part C - Inter-rater Agreement for [68Ga]Ga-DOTA-peptide Per Anatomic Region Between All 4 Raters
Number analyzed (Participants) | 45 | 45
Percentage of Agreement
  Head & Neck | 97.4 | 97.8
  Lung | 97.8 | 98.9
  Liver | 94.4 | 98.5
  Pancreas | 89.3 | 91.5
  Abdomen/Pelvis | 88.5 | 95.2
  Bone | 98.5 | 100
  Lymph Node | 97.4 | 96.3

ADVERSE EVENTS:
Time Frame: Safety data will be collected at baseline and after the administration of the radiotracer for up to 24 hours.
Groups:
- Part A: Patients with histologically-confirmed neuroendocrine tumours (NET) enrolled into Part A of the FETONET study underwent whole-body dynamic [18F]-FET-βAG-TOCA PET/CT imaging at multiple time points over a 4 hour period, with sampling of venous bloods for radioactivity and radioactive metabolite quantification.
- Part B: Patients with histologically confirmed neuroendocrine tumours (NET) underwent PET/CT imaging with both [18F]-FET-βAG-TOCA and [68Ga]Ga-peptide. The two PET/CT scans were performed within a 6-month time period.
  Whole-body static [18F]-FET-βAG-TOCA PET-CT imaging was conducted 50 minutes post-injection.
Arm/Group | Part A | Part B
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/47
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/47
Other Adverse Events (participants affected / at risk) | 2/9 | 1/47
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A (N=9) | Part B (N=47)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypertension (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Altered Taste Sensation (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-12-12): https://cdn.clinicaltrials.gov/large-docs/23/NCT06456723/Prot_SAP_000.pdf